CLINICAL TRIAL: NCT05106348
Title: Methods of Assessing Fitness and Physical Capacity of People With Special Needs - Searching for Guidelines and Methods for Measuring the Population of People With Impairments
Brief Title: Methods of Assessing Fitness and Physical Capacity
Status: Completed | Type: Observational
Sponsor: Jolanta Marszałek (Other)
Collaborators: Polish Wheelchair Rugby Federation (Unknown)
Responsible Party: Sponsor-Investigator, Jolanta Marszałek, associate professor, Józef Piłsudski University of Physical Education
Organization: Józef Piłsudski University of Physical Education (Other)
Other Study IDs: SKE 01-01/2020 (1)
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-10

CONDITIONS: Physical Fitness
Keywords: Capacity; Aerobic Fitness; Protocol; Wheelchair Rugby; Impairments

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wheelchair Rugby Group: wheelchair rugby players, elite athletes, national team athletes
  Interventions: Diagnostic Test: Aerobic Fitness Test

INTERVENTIONS:
Diagnostic Test: Aerobic Fitness Test — aerobic fitness test to assess wheelchair rugby players capacity

SUMMARY:
Aerobic fitness is an important part of sport training preparation for wheelchair rugby players. Currently, there are some test protocols on arm crank ergometer for spinal cord injury people. However, wheelchair propulsion seems to be better and more specific movement to assess aerobic fitness in wheelchair rugby player. Thus, this pilot study was designed to determine the reliability of the aerobic fitness test protocol on a wheelchair ergometer for wheelchair rugby players.

Methods Ten wheelchair rugby players (C5/6 = 4, C6/C7 = 3, C7/th1 = 1 all with incomplete lesions, cerebral palsy (CP) = 1; dysmelia = 1; mean age = 32,90 yr. ± 5,17; body mass = 70,04 kg ± 12,53; body height = 177,70 cm ± 18,64) participated in the aerobic fitness test on the Lode Esseda wheelchair ergometer (LEM Software 10.12, Groningen, Netherlands). This test involved different considering players' International Wheelchair Rugby Federation (IWRF) class (class 0.5 = 4 players, classes 1.0-1.5 = 6 players, and classes 2.0-3.5 = 8 players) increments of workload every minute at constant velocity of 4.5 km/h. Peak oxygen uptake (V̇O2peak l/min, V̇O2peak ml/kg/min), minute ventilation (VE), and the test time achieved were collected (Cortex Metamax). The load [N, Watts] from the last fully achieved level in the test was noticed. Participants repeated the aerobic fitness test twice with 24h break. Each player had 10 minutes warm-up before the test. Differences (T-test for independent groups or Wilcoxon test) and correlations (Pearson test or Spearman test) between results from the first and the second repetition of the test (fully achieved load level in the test) were calculated to establish reliability. The intra-class correlation coefficients (ICC) and standard error of measurement (SEM) were added. The significance level was set at p<.05

DETAILED DESCRIPTION:
"the Lode Esseda" is the name of a wheelchair ergometer.

ELIGIBILITY:
Inclusion Criteria:

- wheelchair rugby players - elite athletes, national team athletes

Exclusion Criteria:

- not healthy participant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: the elite wheelchair rugby players (Polish National Team players) group is a small group of population
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
aerobic fitness test | 13.03.2020-30.06.2021
  Determination the reliability of the aerobic fitness test protocol on a wheelchair ergometer for wheelchair rugby players.

CONTACTS AND LOCATIONS:
Locations (1):
- Jozef Pilsudski University of Physical Education in Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided